CLINICAL TRIAL: NCT05773430
Title: Reducing Cognitive Intra-Individual Variability and Cognitive Impairment in Adults With HIV (The Targeted Neurocognitive Training (TNT) Study)
Brief Title: The Targeted Neurocognitive Training (TNT) Study
Acronym: TNT
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: It got a great score and it looked like it would be funded, but it was never funded.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, David Vance, PhD, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-300010567; UAB (Other: University of Alabama at Birmingham)
Record Dates: First submitted 2023-03-06; First posted 2023-03-17 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: HIV; Aging; Cognitive Function Abnormal; Cognitive Training; Older Adults
Keywords: HIV-Associated Neurocognitive Disorder; cognitive training; executive dysfunction; feasibility
MeSH Terms: conditions — Cognition Disorders

STUDY DESIGN:
Intervention Model Description: A pre-post two-group experimental design will be used. One group will receive the experimental targeted neurocognitive training and the other group will not receive anything (no-contact control group)
Who Masked: Investigator
Masking Description: Testers will be unaware of which training condition participants are assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Targeted Neurocognitive Training (Experimental): BrainHQ (POSIT Science Inc.) computerized cognitive training modules will be used as in our other studies; but these will focus on the two cognitive domains in which the participants exhibited the worst performance at baseline. Twenty hours or training will administer to each participant target these two cognitive domains (10 hours each). These programs have gaming components that encourage adherence. BrainHQ cognitive training products are tested and endorsed by the scientific community. A meta-analysis of computerized cognitive training in older adults found optimal therapeutic effects occurred when training sessions last at most 60 minutes and are administered 1-3 times per week - dosage parameters already incorporated in our study. This self-administered program uses touch-screen technology with tablets which allows computer novices to engage with the training exercises.
  Interventions: Behavioral: Targeted Neurocognitive Training
- No-Contact Control Group (No Intervention): These participants will not receive any intervention.

INTERVENTIONS:
Behavioral: Targeted Neurocognitive Training — Only two cognitive domains will be targeted for training (10 hrs of training in each, for a total of 20 hours). Two or more cognitive exercises may be employed within a cognitive domain. These exercises provide both immediate and intermittent feedback and are customized to the participants' individual ability; the difficulty and/or complexity of each game are systematically decreased/increased based on participants' performance to always be challenging, but not overly frustrating. Typically, in an hour session, one exercise (e.g., Mental Map) will be engaged at a time (20-30 minutes) before switching to another exercise (e.g., Hawkeye) in another domain for 20-30 minutes. This helps the participant remain engaged but avoid fatigue.
  Arms: Targeted Neurocognitive Training

SUMMARY:
People with HIV (PWH) often suffer from cognitive impairments known as HIV-Associated Neurocognitive Disorder (HAND). Cognitive impairments in PWH are not fully captured by traditional neurocognitive assessment; thus, we must examine cognitive performance both within a task (inconsistency) and across cognitive domains (dispersion), called Intra-Individual Variability (IIV). IIV predicts cognitive impairment/decline, altered brain morphology, and neuropathology in many clinical populations. Conceptually, IIV results from "executive dyscontrol" or the efficiency (or inefficiency) with which executive control processes coordinate other cognitive processes/domains. Based on the Executive Dyscontrol Hypothesis and underlying calculations of IIV, one way to improve cognition in PWH is through interventions that target improvements in their most severely impaired cognitive domains. We hypothesize such improvements, in turn, should reduce the strain placed on executive functioning resources, freeing up resources needed to compensate for impairments in any domain and, in turn, reducing IIV. Computerized cognitive training, widely used in the study team's prior work, is ideally suited to target impairments in select cognitive domains using computerized cognitive training. In our systematic review of 13 cognitive training studies in PWH, we found cognitive training improved performance in the targeted domain. In this feasibility study, we will assess 150 PWH at baseline with the expectation to recruit 120 PWH with HAND. Then we will use a two-group pre-post experimental design of 120 adults with HAND including: 1) a Targeted Neurocognitive Training (TNT) group (n=60) to train each participant's two most impaired cognitive domains (e.g., attention & memory) assessed from a neurocognitive battery at baseline, and 2) a no-contact control group (n=60). Aim 1 - Feasibility: To determine feasibility and acceptability of the intervention. Exploratory Aim 1 - Cognition: Compare adults who receive TNT to those who receive no training to determine whether they improve on the cognitive domains trained, show less cognitive IIV across domains and within a task, and demonstrate improved executive functioning. Exploratory Hypothesis 1: TNT will improve cognitive functioning in the targeted impaired cognitive domains. Exploratory Hypothesis 2: TNT will reduce cognitive IIV (both overall dispersion & inconsistency). Exploratory Hypothesis 3: TNT will improve executive functioning. Exploratory Hypothesis 4: TNT will improve global cognition and reduce HAND severity. Innovation 1 - This is the first study to use IIV to guide cognitive training to target the most impaired cognitive domains to reduce cognitive IIV in HIV. Innovation 2 - This will be one of the first studies to prospectively include both types of cognitive IIV - dispersion and inconsistency - allowing us to examine the relationship between dispersion and inconsistency. Innovation 3 - The epicenter of HIV is in the Deep South where this study will occur.

DETAILED DESCRIPTION:
OVERALL -- A pre-post twoe-group experimental design will be used. Participants will be recruited from the University of Alabama at Birmingham (UAB) 1917 HIV/AIDS Clinic which has a patient population of +3,600 and is the largest HIV medical provider within 100 miles. Eligible participants will be consented at the UAB Center for Research on Applied Gerontology where a ~2 hr baseline assessment will be administered. Participants' neuropsychological data gathered at baseline will be examined to determine a HAND classification. Only participants with HIV-Associated Neurocognitive Disorder (HAND) will be invited to continue with the study. Stratified random assignment will ensure an equal number of participants in each group by gender, minority status, and with/without executive functioning impairment (i.e., 1 standard deviation below normative mean). After training, participants will complete a posttest assessment.

Recruitment/Retention Strategies. As effective in our studies, recruitment/retention strategies will be used. 1) Recruitment materials distributed in the UAB 1917 HIV/AIDS Clinic. 2) Reminder letters and telephone calls will be used before the scheduled visit. 3) Beverages/snacks will be provided (from departmental funds). 5) Secondary contact information will be collected to follow up with lost participants.

Intervention Protocol BrainHQ (POSIT Science Inc.) cognitive training modules will be used as in our other studies; these programs have gaming components that encourage adherence. BrainHQ cognitive training products are tested and endorsed by the scientific community. A meta-analysis of computerized cognitive training in older adults found optimal therapeutic effects occurred when training sessions last at most 60 minutes and are administered 1-3 times per week - dosage parameters already incorporated in our study. This self-administered program uses touch-screen technology with tablets which allows computer novices to engage with the training exercises. The intervention will be administered in the research lab of the UAB Center for Applied Gerontology where many of our other studies have been conducted. Working with BrainHQ, when logging on, participants can only receive the individualized cognitive training exercises they are assigned.

Executive Functioning Training Group. Those in the Executive Functioning Training Group will engage in exercises requiring one to set shift; that is, to maintain at least two sets of rules and decide which is appropriate to determine the response. In using these training exercises in the Training On Purpose Study (TOPS), the effects size was quite large (d=-0.89). Dosage of 20 hours of training is considered an upper range on how much training is needed to produce an optimal therapeutic effect.

Targeted Neurocognitive Training (TNT) Group. Only two cognitive domains will be targeted for training (10 hrs of training in each, for a total of 20 hours). Two or more cognitive exercises may be employed within a cognitive domain. These exercises provide both immediate and intermittent feedback and are customized to the participants' individual ability; the difficulty and/or complexity of each game are systematically decreased/increased based on participants' performance to always be challenging, but not overly frustrating. Typically, in an hour session, one exercise (e.g., Mental Map) will be engaged at a time (20-30 minutes) before switching to another exercise (e.g., Hawkeye) in another domain for 20-30 minutes. This helps the participant remain engaged but avoid fatigue.

No-Contact Control Group. This group will receive no intervention. As this is a pilot/feasibility study, investigators do not have the resources to provide a contact control group. Importantly, in a prior study, investigators established that a no-contact control group and a contact control (sham) group did not significantly differ from each other and both served as an excellent comparison to a cognitive intervention.

Instruments Administration time of the assessment will be ~2 hrs. Investigators will use REDCap and BrainBaseline Assessment of Cognition and Everyday Functioning (BRACE+) tablet for administration of the instruments below to reduce tester burden, tester error, and improve the efficiency of data entry and data management, which will save significant staff time and resources. Other cognitive studies as observed in the HIV Neurobehavioral Research Center (HNRC) group employ testing assessments of similar length. BRACE+ was develop in conjunction with HNRC.

ELIGIBILITY:
Inclusion Criteria:

* Participants (men & women) must be 40+ years
* English speaking,
* Have HIV-Associated Neurocognitive Disorder (HAND)
* Willing to meet in person
* Has time to participate for ~12 weeks

Exclusion Criteria:

* Participants living beyond 60 miles away from the center
* Participants living in unstable housing (e.g., halfway house)
* Participants with significant neuromedical comorbidities (e.g., schizophrenia)
* Participants with other conditions (e.g., legally blind/deaf, currently undergoing radiation or chemotherapy, or a history of significant brain trauma, diagnosed with COVID-19 over the past 3 months) that could impact cognitive functioning or testing.
* Participants who have received cognitive training within the past three years- -

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Baseline Assessment of Cognitive Training | ~12 weeks
  All participants at baseline will be asked questions about computer use, knowledge about cognitive training, their perceptions about whether they need cognitive training, knowledge about HIV and cognition, etc. Both quantitative and qualitative (i.e., open-ended responses) data will be collected; this is similar to our other studies
Cognitive Training Satisfaction Questionnaire | ~12 weeks
  Used to assess likes/dislikes of the intervention, both quantitative questions and qualitative (i.e., open-ended responses) data are gathered as has been used in our previous cognitive intervention studies to evaluate feasibility and acceptability.
Exit Survey | ~12 weeks
  Investigators will administer a brief quantitative and qualitative (i.e., open-ended responses) survey to assess what he/she liked/disliked about the training and how to improve it.
Adherence Rates (after study data collection) | Through study completion, an average of 2 years
  Investigators will calculate the adherence rate of the protocol, similar to the investigator's other studies. Ranges will be from 0% to 100%.
Attrition Rates (after study data collection) | Through study completion, an average of 2 years
  Investigators will calculate the attrition rate of the protocol, similar to the investigator's other studies. Ranges will be from 0% to 100%.

SECONDARY OUTCOMES:
BRACE+ (BrainBaseline Assessment of Cognition and Everyday Functioning) | ~12 weeks
  Cognitive data will be gathered via BRACE+ (BrainBaseline Assessment of Cognition and Everyday Functioning), supported by NIMH R42099964 and Digital Artefacts/UCSD) is a HIPAA compliant tablet-based cognitive assessment platform. This self-administered tool is not literacy dependent (i.e., automated audio/video instructions) and uses validated cognitive tests sensitive to mild-to-moderate cognitive impairments.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
We will archive all data electronically without PHI which will be available upon request.
Supporting Information: Study Protocol, SAP
Time Frame: Upon completion of the study
Access Criteria: Based upon IRB approval and Data Use Agreement

REFERENCES:
- [Background] Vance DE, Fazeli PL, Cheatwood J, Nicholson C, Morrison S, Moneyham LD. Targeting HIV-Related Neurocognitive Impairments with Cognitive Training Strategies: Insights from the Cognitive Aging Literature. Curr Top Behav Neurosci. 2021;50:503-515. doi: 10.1007/7854_2018_80. PMID 30710223
- [Background] Vance DE, Fazeli PL, Azuero A, Wadley VG, Raper JL, Ball KK. Can Individualized-Targeted Computerized Cognitive Training Benefit Adults with HIV-Associated Neurocognitive Disorder? The Training on Purpose Study (TOPS). AIDS Behav. 2021 Dec;25(12):3898-3908. doi: 10.1007/s10461-021-03230-y. Epub 2021 Mar 18. PMID 33733311
- [Background] Waldrop D, Irwin C, Nicholson WC, Lee CA, Webel A, Fazeli PL, Vance DE. The Intersection of Cognitive Ability and HIV: A Review of the State of the Nursing Science. J Assoc Nurses AIDS Care. 2021 May-Jun 01;32(3):306-321. doi: 10.1097/JNC.0000000000000232. PMID 33449578